CLINICAL TRIAL: NCT06984406
Title: Randomized Controlled Trial on the Efficacy and Safety of a Beet-Derived Inorganic Nitrate-Based Food Product for the Prevention of Contrast-Induced Nephropathy in High-Risk Patients Undergoing Percutaneous Coronary Intervention (BEET-CIN Trial)
Brief Title: Efficacy and Safety of a Beet-Derived Inorganic Nitrate-Based Food Product for the Prevention of Contrast-Induced Nephropathy in High-Risk Patients Undergoing Percutaneous Coronary Intervention
Acronym: BEET-CIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-02/25
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Contrast-induced Nephropathy Following Percutaneous Intervention (CIN)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate Supplementation Group (Experimental): Participants in this arm will receive standard preventive measures for contrast-induced nephropathy, including adequate hydration and contrast volume minimization and in addition beet-derived inorganic nitrate-based food product as an oral supplement for 5 days. The intervention will start 24 hours before PCI and continue for 4 days post-procedure. The supplementation aims to enhance renal perfusion, reduce oxidative stress, and prevent contrast-induced nephropathy.
  Interventions: Dietary Supplement: Beet-Derived Inorganic Nitrate-Based Food Product
- Standard Care Group (No Intervention): Participants in this arm will receive standard preventive measures for contrast-induced nephropathy, including adequate hydration and contrast volume minimization, but will not receive the nitrate-based supplement.

INTERVENTIONS:
Dietary Supplement: Beet-Derived Inorganic Nitrate-Based Food Product — This intervention consists of an orally administered food product enriched with inorganic nitrates derived from beetroot. Participants in the intervention group will consume a standardized dose of 12 mmol of nitrate per day for 5 days (starting 24 hours before PCI and continuing for 4 days post-procedure). The product is designed to enhance nitric oxide bioavailability, improve renal perfusion, reduce oxidative stress, and lower the risk of contrast-induced nephropathy (CIN).
  Arms: Nitrate Supplementation Group

SUMMARY:
Contrast-induced nephropathy (CIN) is a common complication in high-risk patients undergoing percutaneous coronary intervention (PCI) due to exposure to iodinated contrast agents. CIN is associated with increased morbidity, prolonged hospital stays, and higher healthcare costs. Current preventive strategies include adequate hydration and minimizing contrast volume; however, there is no universally effective pharmacological intervention.

Recent studies suggest that inorganic nitrates can enhance renal perfusion, reduce oxidative stress, and improve endothelial function, potentially lowering the risk of CIN. This study aims to evaluate the efficacy and safety of a beet-derived inorganic nitrate-based food product for the prevention of CIN in high-risk patients undergoing PCI.

This is a randomized, controlled, open-label clinical trial comparing two groups:

1. Intervention Group: Patients receiving the beet-derived inorganic nitrate-based food product for 5 days (starting 24 hours before PCI).
2. Control Group: Patients receiving standard medical care without additional nitrate supplementation.

We hypothesize that the nitrate-based food product will significantly reduce the incidence of CIN compared to standard care. Additionally, we expect:

1. A lower increase in kidney injury biomarkers (NGAL, cystatin C) in the intervention group.
2. A slower decline or even improvement in eGFR at follow-up.
3. A potential reduction in MACE due to the vasoprotective effects of nitrates.
4. Improved quality of life scores (EQ-5D) in the intervention group. If successful, this study will provide new evidence supporting the use of dietary nitrates for renal protection and may contribute to the development of novel, cost-effective prevention strategies for CIN.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Planned PCI.
* High risk of CIN with:

  1. eGFR according to the CKD-EPI formula <60 ml/min/1.73 m2 or
  2. At least two of the following criteria: liver damage (cirrhosis), diabetes mellitus, age >70 years, administration of contrast in the last 7 days, CHF (LVEF >40%), intake of drugs affecting renal function (ACE inhibitors, ARBs, NSAIDs, aminoglycosides, diuretics).
* Signing informed consent.

Exclusion Criteria:

* Allergy to nitrates.
* Acute coronary syndrome.
* Acute condition accompanied by systolic blood pressure <90 mmHg for more th an 30 minutes or requiring the use of drugs with a positive inotropic effect.
* Life-threatening conditions requiring emergency medical care.
* Participation in other clinical trials.
* Pregnancy, lactation.
* Use of nitrates in the last 30 days.
* Abuse of alcohol, illegal drugs, mnestic-intellectual decline, as well as other reasons and circumstances indicating expected low adherence to treatment.
* Refusal to follow the plan of visits and examinations provided for by the protocol of this clinical trial.
* Refusal to sign informed consent.
* Infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Contrast-Induced Nephropathy (CIN) | Baseline, 48 hours post-PCI
  Contrast-induced nephropathy (CIN) will be defined based on KDIGO criteria as:
  * An increase in serum creatinine of ≥0.3 mg/dL (26.52 μmol/L) within 48 hours post-PCI, OR
  * An increase in serum creatinine of ≥1.5 times from baseline within 7 days post-PCI.
  * A urine output < 0.5 mL/kg/hour for six hours. The incidence of CIN will be compared between the intervention (nitrate supplementation) and control groups.

SECONDARY OUTCOMES:
Changes in Renal Function Biomarkers (NGAL, Cystatin C, eGFR) | Baseline, 4-6 hours, 24 hours, 48 hours, and 3 months post-PCI
  Neutrophil gelatinase-associated lipocalin (NGAL) and Cystatin C will be measured at baseline, 4-6 hours, 24 hours, and 48-72 hours post-PCI to assess early kidney injury.
  Estimated glomerular filtration rate (eGFR) will be calculated at baseline, 48-72 hours, and 3 months post-PCI to evaluate long-term renal function changes.
Incidence of Major Adverse Cardiovascular Events (MACE) | 3 months and 12 months post-PCI
  MACE will be defined as the composite of:
  Cardiovascular death
  Myocardial infarction
  Stroke
  Unplanned coronary revascularization The incidence will be compared between the two study arms.
Quality of Life Assessment (EQ-5D Score) | Baseline and 12 months post-PCI
  Changes in quality of life will be assessed using the EQ-5D questionnaire, a validated tool measuring five dimensions:
  Mobility
  Self-care
  Usual activities
  Pain/discomfort
  Anxiety/depression Scores will be compared between groups to evaluate the impact of nitrate supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution National Medical Research Center for Therapy and Preventive Medicine of the Ministry of Healthсare of the Russian Federation, Moscow, Russia